CLINICAL TRIAL: NCT04520932
Title: Pancreatic Radiofrequency Under High Echo-endoscopy in the Management of Low Grade Pancreatic Neuroendocrine Tumors of Less Than 2cm in Size
Brief Title: Pancreatic Radiofrequency Under High Echo-endoscopy in the Management of Pancreatic Neuroendocrine Tumors
Acronym: RFANET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFANET-IPC 2020-003
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumor of Pancreas (Disorder); Neuroendocrine Tumor Grade 1
Keywords: Radio Frequency treatment; Echoendoscopy; Ablation; Efficacy
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA treatment efficacy (Experimental): PNETs ablation by radiofrequency treatment (1 to 3 sessions)
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — RFA is performed under general anaesthesia, under high endoscopic echo-endoscopy (EEH), in left lateral decubitus position, using the StarMed generator from Taewong®.

SUMMARY:
Pancreatic radiofrequency ablation (RFA) could therefore be an alternative to the monitoring of pancreatic neuroendocrine tumors (PNETs) and more particularly nonfunctioning PNETs (NF-PNETs), which is costly and anxiety-inducing for patients. To date, only a few small studies have evaluated this treatment and the results are encouraging. It appears necessary to consider a large-scale study to ensure the efficacy and low morbidity of pancreatic RFA applied to PNETs.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of radiofrequency treatment of grade 1 NF-PNETS with a size less than or equal to 2cm.

Patients meeting the selection criteria will be included in the study after signing the consent. They will benefit from a RFA treatment consisting of 1 to 3 sessions depending on their response to the treatment. Patients will then be followed for 5 years in order to evaluate their response to treatment, their clinical evolution, their quality of life and any complications.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic mass of less than 2cm on MRI, or CT scan if contraindicated by MRI;
* Diagnosis of neuroendocrine tumor on biopsy under high echo-endoscopy (HEE) with Ki67<3%,
* Non-secretory lesion.
* Homogeneous HEE contrast taking;
* No positron emission tomography (PET) FDG binding to the pancreatic mass;
* Lesion <20mm on conventional imaging at 6 months monitoring;
* Age 18 to 80 years inclusive;
* Patient in good general condition, World Health Organization [0-1];
* Signed consent to participate;
* Affiliation to healthcare insurance system or beneficiary of this regimen.

Exclusion Criteria:

* Pregnant or likely to become pregnant (without effective contraception) or breastfeeding ;
* A person in an emergency situation or deprived of liberty or placed under the authority of a tutor.
* Life expectancy < 1 year;
* Severe hemostasis disorders;
* Pancreatic and/or biliary ductal dilation;
* Lesion considered to be adjacent to the pancreatic duct and/or bile duct;
* Node extension and/or metastatic disease;
* Patient being managed for another malignant lesion which is progressive or under treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Treatment response | 1 year
  Complete response rate to radiofrequency treatment defined by the absence of enhancement with the contrast agent and/or the disappearance of the lesion on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice CAILLOL, MD, Principal Investigator — Paoli Calmettes Institute
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No